CLINICAL TRIAL: NCT05918666
Title: National Register of Actionable Mutations - Rational Study
Brief Title: National Register of Actionable Mutations
Acronym: RATIONAL
Status: Active, not recruiting | Type: Observational
Sponsor: Federation of Italian Cooperative Oncology Groups (Other)
Collaborators: Roche Pharma AG (Industry); AstraZeneca (Industry); Bayer (Industry); Bristol-Myers Squibb (Industry); Janssen, LP (Industry); Takeda (Industry); Amgen (Industry); Daiichi Sankyo (Industry); Eli Lilly and Company (Industry); Novartis (Industry); Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: Rational study
Record Dates: First submitted 2023-05-30; First posted 2023-06-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumours in Advanced Stages

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is the creation of a national network of precision medicine, which allows to increase, for Italian patients suffering from solid tumors, the possibility of access to more innovative therapies and to collect retrospectively their clinical data.

For this purpose, a national register of actionable mutations in patients with solid tumors in advanced stage of disease will be created in which various individual, local and regional initiatives of genomic screening of cancer could merge.

DETAILED DESCRIPTION:
The primary objective of this observational study is to describe the frequency of actionable mutations in patients with solid tumors in advanced stage, receiving a genetic-molecular characterization with high throughput methods.

The secondary objectives are:

1. assess the correlation between genetic alterations and clinical and pathological characteristics of enrolled patients (gender, age, histological variant, location and extent of neoplasm, comorbidity, familiarity for neoplasms);
2. describe, where possible, any variation in the molecular profile for patients who are subjected to genetic screening analysis at different stages of the disease.
3. record retrospectively clinical efficacy and toxicity data when patients were treated with a target therapy based on the detected molecular alterations.

The national register of actionable mutations will be created collecting the following data:

1. Data extracted retrospectively from medical records of patients that have received during the study period a test with high-throughput technologies for the molecular characterization of their tumor, either by clinical routine or for research purposes.
2. Data collected prospectively from analysis of biological samples (FFPE and biopsy liquid) of patients that meet the elibility criteria and that perform the molecular-genetic screening using Foundation Medicine services or in selected italian laboratories.
3. Clinical data collected retrospectively (RR, DOR, PFS, OS, toxicity), in case where the patients are treated with a target therapy, based on the highlighted molecular alterations and on the choice of the clinician.

Only samples already available for clinical practice will be used in the study.

The register will be limited to collecting information on molecular alterations that can then be used for the insertion of patients in clinical studies already active, for the design of new studies proposed by members of the Steering Committee or of the participating sites, or for treatment with other modality.

ELIGIBILITY:
General Inclusion Criteria for all patients:

* Age >18 years old
* Life expectancy 6 months
* ECOG performance status 2
* Diagnosis of malignant solid tumor, in advanced stage
* Informed consent to data registration and for privacy purposes

Additional inclusion criteria for patients that have already carried out a genetic characterisation extended by high throughput methods:

● Availability of the result of the broad spectrum analysis of genetic alterations carried out with high throughput methods on biological samples

Additional inclusion criteria for patients that perform the molecular-genetic screening using Foundation Medicine services or in selected italian laboratories:

* one of the following criteria:

  * Patients diagnosed with NSCLC not squamous, not pretreated;
  * Patients with biliary tract, pancreatic, esophagus, stomach, thymus, CNS, nasopharynx, salivary glands, endometrium and urothelium cancers;
  * Patients with any disease (including NSCLC) who are progressing disease after treatment with molecular target drugs. For these patients is the availability of a post- treatment biological sample is necessary;
  * Patients with cancer of unknown primary (CUP);
  * Young patients (<40 years) or patients who have exhausted standard lines of therapy, with any advanced/metastatic tumor which, in the opinion of the investigator, may benefit from a genetic-molecular characterization at broad spectrum aimed at a treatment with molecular target therapies.
* availability of biological material for testing.
* informed consent for testing.

Additional exclusion criteria for patients that perform the molecular-genetic screening using Foundation Medicine services or in selected italian laboratories:

● patients who have already received NGS or other high throughput in the same stage of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with solid tumors in advanced stage of disease
Sampling Method: Probability Sample
Enrollment: 2098 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
rate of actionable mutations identified with NGS | from October 2018 to study completion, 2 years after the last enrolled patient
  information on somatic mutations obtained by analysis of neoplastic tissue samples and/or liquid biopsy (circulating tumor DNA extracted from the patient's plasma).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Normanno, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori S.r.l. IRCCS
Locations (43):
- Italy (43):
  - S.O.D. Clinica Oncologica - A.O.U. Ospedali Riuniti Ancona, Ancona
  - U.O.C. Oncologia Medica - Ospedale San Donato, Arezzo
  - U.O. Oncologia Medica - A.O. S.G. Moscati, Avellino
  - Divisione di Oncologia Medica e dei Tumori Immunocorrelati - Centro di Riferimento Oncologico, Aviano
  - U.O.C. Oncologia Medica e Sperimentale - Istituto Tumori Giovanni Paolo II IRCCS, Bari
  - U.O. Oncologia Medica - Humanitas Gavazzeni, Bergamo
  - Unità di Struttura Complessa Oncologia Medica - ASST Papa Giovanni XXIII, Bergamo
  - Oncologia Medica e Brest Unt - Presidio di Brindisi Di Summa-Perrino, Brindisi
  - U.O.C. Oncologia Medica - A.O.U. Policlinico Vittorio Emanuele, Catania
  - U.O.C. Oncologia Medica - Ospedale Garibaldi Nesima, Catania
  - S.C. di Oncologia Medica - A.O.U. Careggi, Florence
  - U.O.S. Tumori polmonari IRCCS A.O.U. San Martino IST - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - U.O. Oncologia Medica - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori S.r.l. IRCCS, Meldola
  - Oncologia - AOU Policlinico "G. Martino", Messina
  - U.O. Oncologia Medica - A.O. Papardo, Messina
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Niguarda Cancer Center - Ospedale Niguarda e Università degli Studi di Milano, Milan
  - Oncologia Toracica - Istituto Europeo di Oncologia, Milan
  - Sviluppo di nuovi Farmaci per Terapie Innovative - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale, Napoli
  - Oncologia Medica - A.O.U. Seconda Università degli studi di Napoli, Napoli
  - U.O.C. Oncologia - AORN - Ospedali dei Colli, Napoli
  - U.O.C. Oncologia - Asl Napoli 1 Centro - Ospedale del Mare, Napoli
  - Oncologia - Ospedale Sacro Cuore Don Calabria, Negrar
  - U.O. Oncologia Medica 2 - Istituto Oncologico Veneto, Padua
  - Oncologia Medica - A.O.U. Policlinico Paolo Giaccone, Palermo
  - S.C. Oncologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - S.C. Oncologia Medica - A.O. S.M. della Misericordia, Perugia
  - U.O. Oncologia Medica 2 - Stabilimenteo S. Chiara - A.O.U. Pisana, Pisa
  - S.C. Oncologia - IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia
  - Day Hospital - Oncologia Medica - Università Campus Biomedico di Roma, Roma
  - U.O.C. Oncologia - A.O. San Camillo -Forlanini, Roma
  - U.O.C. Oncologia - A.O. Sant'Andrea, Roma
  - U.O.S.D. Pneumologia Oncologica - San Camillo Forlanini, Roma
  - U.O.C. Oncologia - A.O.U. OO.RR. San Giovanni di Dio Ruggi d'Aragona, Salerno
  - S.C. Oncologia - Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Dipartimento di Oncologia - A.O.U. San Luigi Gonzaga, Torino
  - S.C. Oncologia - Ospedale Humanitas Gradenigo, Torino
  - U.O. Oncologia Medica - Ospedale Santa Chiara, Trento
  - U.O.C. Oncologia - ASST Bergamo ovest, Treviglio
  - UOC Oncologia Medica - ULSS 2 Marca Trevigiana - P.O. Treviso, Treviso
  - Dipartimento ad attività integrata di Oncologia - Azienda Sanitaria Universitaria Integrata di Udine Friuli Centrale, Udine
  - U.O.C. di Oncologia medica - A.O.U. Integrata Verona, Verona

REFERENCES:
- [Background] Barlesi F, Mazieres J, Merlio JP, Debieuvre D, Mosser J, Lena H, Ouafik L, Besse B, Rouquette I, Westeel V, Escande F, Monnet I, Lemoine A, Veillon R, Blons H, Audigier-Valette C, Bringuier PP, Lamy R, Beau-Faller M, Pujol JL, Sabourin JC, Penault-Llorca F, Denis MG, Lantuejoul S, Morin F, Tran Q, Missy P, Langlais A, Milleron B, Cadranel J, Soria JC, Zalcman G; Biomarkers France contributors. Routine molecular profiling of patients with advanced non-small-cell lung cancer: results of a 1-year nationwide programme of the French Cooperative Thoracic Intergroup (IFCT). Lancet. 2016 Apr 2;387(10026):1415-1426. doi: 10.1016/S0140-6736(16)00004-0. Epub 2016 Jan 15. PMID 26777916
- [Background] Burrell RA, Swanton C. Tumour heterogeneity and the evolution of polyclonal drug resistance. Mol Oncol. 2014 Sep 12;8(6):1095-111. doi: 10.1016/j.molonc.2014.06.005. Epub 2014 Jul 10. PMID 25087573
- [Background] Davis W, Makar G, Mehta P, Zhu GG, Somer R, Morrison J, Kubicek GJ. Next-Generation Sequencing in 305 Consecutive Patients: Clinical Outcomes and Management Changes. J Oncol Pract. 2019 Dec;15(12):e1028-e1034. doi: 10.1200/JOP.19.00269. Epub 2019 Aug 2. PMID 31373836
- [Background] Garraway LA. Genomics-driven oncology: framework for an emerging paradigm. J Clin Oncol. 2013 May 20;31(15):1806-14. doi: 10.1200/JCO.2012.46.8934. Epub 2013 Apr 15. PMID 23589557
- [Background] Kris MG, Johnson BE, Berry LD, Kwiatkowski DJ, Iafrate AJ, Wistuba II, Varella-Garcia M, Franklin WA, Aronson SL, Su PF, Shyr Y, Camidge DR, Sequist LV, Glisson BS, Khuri FR, Garon EB, Pao W, Rudin C, Schiller J, Haura EB, Socinski M, Shirai K, Chen H, Giaccone G, Ladanyi M, Kugler K, Minna JD, Bunn PA. Using multiplexed assays of oncogenic drivers in lung cancers to select targeted drugs. JAMA. 2014 May 21;311(19):1998-2006. doi: 10.1001/jama.2014.3741. PMID 24846037
- [Background] Lopez-Chavez A, Thomas A, Rajan A, Raffeld M, Morrow B, Kelly R, Carter CA, Guha U, Killian K, Lau CC, Abdullaev Z, Xi L, Pack S, Meltzer PS, Corless CL, Sandler A, Beadling C, Warrick A, Liewehr DJ, Steinberg SM, Berman A, Doyle A, Szabo E, Wang Y, Giaccone G. Molecular profiling and targeted therapy for advanced thoracic malignancies: a biomarker-derived, multiarm, multihistology phase II basket trial. J Clin Oncol. 2015 Mar 20;33(9):1000-7. doi: 10.1200/JCO.2014.58.2007. Epub 2015 Feb 9. PMID 25667274
- [Background] Meric-Bernstam F, Brusco L, Shaw K, Horombe C, Kopetz S, Davies MA, Routbort M, Piha-Paul SA, Janku F, Ueno N, Hong D, De Groot J, Ravi V, Li Y, Luthra R, Patel K, Broaddus R, Mendelsohn J, Mills GB. Feasibility of Large-Scale Genomic Testing to Facilitate Enrollment Onto Genomically Matched Clinical Trials. J Clin Oncol. 2015 Sep 1;33(25):2753-62. doi: 10.1200/JCO.2014.60.4165. Epub 2015 May 26. PMID 26014291
- [Background] Normanno N, Rachiglio AM, Roma C, Fenizia F, Esposito C, Pasquale R, La Porta ML, Iannaccone A, Micheli F, Santangelo M, Bergantino F, Costantini S, De Luca A. Molecular diagnostics and personalized medicine in oncology: challenges and opportunities. J Cell Biochem. 2013 Mar;114(3):514-24. doi: 10.1002/jcb.24401. PMID 22991232
- [Background] Pishvaian MJ, Blais EM, Brody JR, Lyons E, DeArbeloa P, Hendifar A, Mikhail S, Chung V, Sahai V, Sohal DPS, Bellakbira S, Thach D, Rahib L, Madhavan S, Matrisian LM, Petricoin EF 3rd. Overall survival in patients with pancreatic cancer receiving matched therapies following molecular profiling: a retrospective analysis of the Know Your Tumor registry trial. Lancet Oncol. 2020 Apr;21(4):508-518. doi: 10.1016/S1470-2045(20)30074-7. Epub 2020 Mar 2. PMID 32135080
- [Background] Smyth LM, Zhou Q, Nguyen B, Yu C, Lepisto EM, Arnedos M, Hasset MJ, Lenoue-Newton ML, Blauvelt N, Dogan S, Micheel CM, Wathoo C, Horlings H, Hudecek J, Gross BE, Kundra R, Sweeney SM, Gao J, Schultz N, Zarski A, Gardos SM, Lee J, Sheffler-Collins S, Park BH, Sawyers CL, Andre F, Levy M, Meric-Bernstam F, Bedard PL, Iasonos A, Schrag D, Hyman DM; AACR Project GENIE Consortium. Characteristics and Outcome of AKT1 E17K-Mutant Breast Cancer Defined through AACR Project GENIE, a Clinicogenomic Registry. Cancer Discov. 2020 Apr;10(4):526-535. doi: 10.1158/2159-8290.CD-19-1209. Epub 2020 Jan 10. PMID 31924700